CLINICAL TRIAL: NCT02547805
Title: A Phase 2, Multicenter, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy and Safety of ALLN-177 Treatment Over 28 Days in Patients With Secondary Hyperoxaluria and Kidney Stones
Brief Title: Evaluate the Effect of ALLN-177 in Reducing Urinary Oxalate in Patients With Secondary Hyperoxaluria and Kidney Stones Over 28 Days
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000713
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Secondary Hyperoxaluria; Nephrolithiasis; Hyperoxaluria; Kidney Stones; Dietary Hyperoxaluria
Keywords: Urine Oxalate; Nephrolithiasis; Kidney Stones; Hyperoxaluria; Enteric Hyperoxaluria; Idiopathic Hyperoxaluria; Urological Diseases; Kidney Diseases; Supersaturation; Dietary Oxalate
MeSH Terms: conditions — Nephrolithiasis; Hyperoxaluria; Kidney Calculi; Urologic Diseases; Kidney Diseases | interventions — reloxaliase; oxalate decarboxylase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Five (5) capsules of placebo by mouth (PO) three times per day (TID) with meals
  Interventions: Drug: Placebo
- ALLN-177 (Experimental): Five (5) capsules of ALLN-177 (1,500 units per capsule) PO TID with meals
  Interventions: Drug: ALLN-177

INTERVENTIONS:
Drug: ALLN-177 — ALLN-177 7,500 units (5 capsules) PO TID with meals
  Other Names: Oxalate decarboxylase
  Arms: ALLN-177
Drug: Placebo — Placebo 5 capsules PO TID with meals
  Arms: Placebo

SUMMARY:
Evaluate the safety, tolerability, and efficacy of 28 days of treatment with ALLN-177 for reducing urinary oxalate excretion in patients with secondary hyperoxaluria and kidney stones.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo controlled study to evaluate the efficacy of ALLN 177 compared with placebo in reducing the urinary excretion of oxalate in subjects with secondary hyperoxaluria and kidney stones. ALLN-177 is an orally administered form of oxalate decarboxylase. The goal of therapy with ALLN-177 is to reduce urinary oxalate excretion by decreasing the absorption of oxalate from the gastrointestinal tract.

Eligible subjects will be randomized to 28 days of treatment with ALLN-177 (7,500 units) or placebo three times daily with meals. Urinary oxalate excretion will be assessed by 24-hr urine collections throughout the study.

The study allows for approximately 66 subjects. The number of enrolled subjects may be increased to a maximum of 100 following an interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* History of enteric or idiopathic hyperoxaluria or kidney stones
* Urinary oxalate ≥ 50 mg/24 hours

Exclusion Criteria:

* Hyperuricosuria
* Glomerular filtration rate < 45 mL/min/1.73m2
* Hypercalcemia or hyperthyroidism
* Autoimmune disorder requiring systemic steroids
* Acute renal colic, primary hyperoxaluria, pure uric acid and/or cysteine stones, renal tubular acidosis, chronic urinary tract infection, or acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mean change in urinary oxalate excretion (mg/24h) | 28 days

SECONDARY OUTCOMES:
Percent change in urinary oxalate excretion | 28 days
≥ 7.5 mg/24 hr decrease in urinary oxalate | 28 days
≥ 10 mg/24 hr decrease in urinary oxalate | 28 days
Mean change in urinary supersaturation of calcium oxalate | 28 days
Time-weighted average urinary oxalate excretion (mg/24h) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Kausz, MD MS, Study Director — VP Clinical Development
Locations (22):
- United States (22):
  - Mayo Clinica Arizona, Pheonix, Arizona
  - Urological Associates of Southern Arizona, PC, Tuscon, Arizona
  - Applied Research Center of Arkansas, Inc., Little Rock, Arkansas
  - South Florida Medical Research, LLC, Aventura, Florida
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Idaho Urological Institute, Meridian, Idaho
  - IU Health Physicians Urology, Indianapolis, Indiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Department of Medicine Clinical Trials Unit, Rochester, Minnesota
  - Delaware Valley Urology, LLC, Voorhees Township, New Jersey
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Coastal Urology, Wilmington, North Carolina
  - Tristate Urologic Services PSC INC. DBA The Urology group, Cincinnati, OH, Ohio
  - Clinical Research Solutions, LLC, Middleburg Heights, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas PLLC, Dallas, Texas
  - Urology of Virginia, Virginia Beach, Virginia
  - Integrity Medical Research, Mountlake Terrace, Washington

IPD SHARING:
Plan to Share IPD: No